CLINICAL TRIAL: NCT00133991
Title: Phase II Study of Intensified CVP, Rituximab, and High Dose Cyclophosphamide for Adult Burkitt or Burkitt-Like Lymphoma
Brief Title: Combination Chemotherapy and Rituximab in Treating Patients With Newly Diagnosed Burkitt's Lymphoma or Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0409; P50CA096888 (NIH); P30CA006973 (NIH); NA_00035765 (Other: JHMIRB)
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Leukemia; Lymphoma
Keywords: untreated adult acute lymphoblastic leukemia; L3 adult acute lymphoblastic leukemia; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma; stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Burkitt Lymphoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Rituximab; Cyclophosphamide; Cytarabine; Methotrexate; Prednisone; Hydrocortisone; Vincristine; Leucovorin

ARMS (1):
- R-CVP + HiCy (Experimental): Protocol intervention consists of two fifteen-day cycles of cyclophosphamide (Cy), vincristine (V), prednisone (P), rituximab (R), with filgrastim support. CNS intervention consists of three days of cytarabine and hydrocortisone and one day of methotrexate (with leucovorin support) for each cycle. After those two cycles, rituximab and high-dose cyclophosphamide (HiCy) will be given.
  Interventions: Biological: Filgrastim; Biological: Rituximab; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Methotrexate; Drug: Prednisone; Drug: Hydrocortisone; Drug: Vincristine; Drug: Leucovorin

INTERVENTIONS:
Biological: Filgrastim — 5 mcg/kg/day starting on Day 3 after each R-CVP cycle and on Day 6 after HiCy.
  Other Names: Neupogen; G-CSF
Biological: Rituximab — 375 mg/m^2 on Day 1 and Day 8 of each R-CVP cycle. 375 mg/m^2 on Day -4 of HiCy and weekly for four weeks after HiCy.
  Other Names: Rituxan
Drug: Cyclophosphamide — 1500 mg/m^2 on Day 1 of each R-CVP cycle. 50 mg/kg/day on Days -3, -2, -1, and 0 of HiCy.
  Other Names: Cytoxan; Cy; CTX; HiCy
Drug: Cytarabine — 100 mg intrathecal on Days 1, 4, and 11 of each cycle of R-CVP.
  Other Names: Ara-C
Drug: Methotrexate — 3 g/m^2 on Day 8 of each cycle of R-CVP.
  Other Names: MTX
Drug: Prednisone — 100 mg on Days 1-5 of each cycle of R-CVP.
  Other Names: Deltasone
Drug: Hydrocortisone — 50 mg intrathecal on Days 1, 4, and 11 of each cycle of R-CVP.
Drug: Vincristine — 1.4 mg/m^2 on Day 1 of each cycle of R-CVP.
  Other Names: Oncovin
Drug: Leucovorin — 25 mg four times daily after methotrexate administration. Dosing continues until adequate methotrexate levels are reached.
  Other Names: Folinic acid

SUMMARY:
RATIONALE: Drugs used in chemotherapy, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving combination chemotherapy together with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with rituximab works in treating patients with newly diagnosed Burkitt's lymphoma or leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall response rate, 1-year event-free survival, and overall survival of adult patients with newly diagnosed Burkitt or atypical Burkitt lymphoma or leukemia treated with dose-intensified induction therapy comprising cyclophosphamide, vincristine, prednisone, and rituximab followed by consolidation therapy comprising rituximab and high-dose cyclophosphamide.
* Determine the grade 3 or higher non-hematologic toxic effects and overall tolerability of this regimen in these patients.

Secondary

* Determine the 3-year event-free survival and overall survival of patients treated with this regimen.
* Determine the general patterns of CNS and systemic relapse in patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Dose-intensified CVP induction therapy: Patients receive cyclophosphamide IV and vincristine IV on day 1. Patients also receive oral prednisone on days 1-5 and rituximab IV on days 1 and 8, and high-dose methotrexate IV with leucovorin calcium IV rescue on day 8. Patients receive filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 3 and continuing until blood counts recover. Treatment repeats approximately every 14 days for 2 courses.
* CNS therapy: Patients receive cytarabine intrathecally (IT) with or without hydrocortisone IT on days 1, 4, and 11 of each induction therapy course. Patients with evidence of CNS involvement by lymphoma continue to receive cytarabine IT twice weekly during any induction therapy treatment delay. Patients who demonstrate CSF clearance receive cytarabine IT once weekly for 4 doses and then once every other week for 4 doses during consolidation therapy. Patients with disease progression during induction therapy or persistent CNS involvement by lymphoma are removed from the study. All other patients proceed to consolidation therapy.
* Consolidation therapy: Patients receive rituximab IV on day -4 and high-dose cyclophosphamide IV on days -3, -2, -1, and 0. Patients receive G-CSF SC once daily beginning on day 6 and continuing until blood counts recover OR pegfilgrastim SC once on day 6. Patients then receive rituximab IV once weekly for 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 3 years.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Classic, sporadic Burkitt's lymphoma
  * Burkitt's leukemia (FAB L3 acute lymphoblastic leukemia)
  * Atypical Burkitt/Burkitt's-like lymphoma or leukemia, defined by the following criteria:

    * Characteristic morphologic features
    * High proliferative index AND Ki-67 ≥ 85%
* Any stage allowed
* Newly diagnosed or untreated disease

  * Steroids allowed

PATIENT CHARACTERISTICS:

Age

* 30 and over

Performance status

* Not specified

Life expectancy

* Not specified

Renal

* No known irreversible renal dysfunction that would preclude treatment with high-dose cyclophosphamide

Cardiovascular

* No known significant cardiac dysfunction that would preclude treatment with high-dose cyclophosphamide

Other

* Not pregnant or nursing
* No known HIV positivity
* No other malignancy within the past 3 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for lymphoma

  * A maximum of 2 prior doses of intrathecal chemotherapy are allowed

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiation therapy for lymphoma

Surgery

* Prior complete or incomplete surgical resection of lymphoma allowed

Ages: 30 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-07 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvette L. Kasamon, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Drexel University College of Medicine - Center City Hahnemann Campus, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kasamon YL, Brodsky RA, Borowitz MJ, Ambinder RF, Crilley PA, Cho SY, Tsai HL, Smith BD, Gladstone DE, Carraway HE, Huff CA, Matsui WH, Bolanos-Meade J, Jones RJ, Swinnen LJ. Brief intensive therapy for older adults with newly diagnosed Burkitt or atypical Burkitt lymphoma/leukemia. Leuk Lymphoma. 2013 Mar;54(3):483-90. doi: 10.3109/10428194.2012.715346. Epub 2012 Aug 17. PMID 22835045

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants were found to be HIV+ after initiating the study and are considered to be screen failures as defined by the protocol.
Period: Overall Study
Arm/Group | R-CVP + HiCy
Started | 21
Completed | 17
Not Completed | 4
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | R-CVP + HiCy
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 53 [34 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Number of participants who have a complete or partial remission (2007 International Working Group criteria).
Time Frame: Up to 3 months
Population: The 4 participants who died during treatment were not analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | R-CVP + HiCy
Number analyzed (Participants) | 17
Participants
  Complete remission | 11
  Partial remission | 2

2. Primary Outcome: Overall Survival
Description: Percentage of participants alive at 1 year and at 3 years.
Time Frame: 1 year and 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-CVP + HiCy
Number analyzed (Participants) | 21
percentage of participants
  1 year | 57 [40 to 83]
  3 years | 57 [40 to 83]

3. Primary Outcome: Event-free Survival
Description: Percentage of participants alive without relapse at 1 year and 3 years.
Time Frame: 1 year and 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-CVP + HiCy
Number analyzed (Participants) | 21
percentage of participants
  1 year | 52 [35 to 79]
  3 years | 52 [35 to 79]

4. Primary Outcome: Percentage of Participants Experiencing Grade 3-5 Toxicity
Description: Percentage of participants experiencing at least one grade 3-5 adverse event (by CTCAE 3.0 criteria).
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | R-CVP + HiCy
Number analyzed (Participants) | 21
Participants | 21

5. Secondary Outcome: Relapse Pattern
Description: Percentage of participants experiencing central nervous system (CNS) and systemic relapse.
Time Frame: Up to 6 months
Population: The 4 participants who died during treatment were not analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | R-CVP + HiCy
Number analyzed (Participants) | 17
Participants
  Systemic relapse only | 3
  Systemic and CNS relapse | 2

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Adverse events were tracked monthly through the completion of study intervention and then every three months for up to two years total.
Arm/Group | R-CVP + HiCy
All-Cause Mortality (participants affected / at risk) | 9/21
Serious Adverse Events (participants affected / at risk) | 12/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-CVP + HiCy (N=21)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ascites (Hepatobiliary disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Blood infection (Infections and infestations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1)
Febrile neutropenia (Infections and infestations) | 2 (2)
Hypotension (Cardiac disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain - chest (Musculoskeletal and connective tissue disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Somnolence (General disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Subdural hematoma (Nervous system disorders) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Wound complication (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-CVP + HiCy (N=21)
Allergic reaction (Immune system disorders) | 3 (3)
Anasarca (General disorders) | 2 (2)
Anemia (Investigations) | 3 (6)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Blurred vision (Nervous system disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (4)
Chills (General disorders) | 3 (5)
Confusion (Nervous system disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 9 (19)
Cough (General disorders) | 3 (5)
Anorexia (Gastrointestinal disorders) | 3 (3)
Deep vein thrombosis (Cardiac disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 6 (12)
Dizziness (Nervous system disorders) | 4 (7)
Drowsiness (Nervous system disorders) | 2 (4)
Dysphagia (Gastrointestinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (18)
Edema (Cardiac disorders) | 5 (10)
Facial droop (Nervous system disorders) | 2 (2)
Fatigue (General disorders) | 7 (13)
Febrile neutropenia (Infections and infestations) | 6 (8)
Fever (Infections and infestations) | 6 (14)
Hallucination (Nervous system disorders) | 2 (3)
Headache (General disorders) | 11 (27)
Hematuria (Renal and urinary disorders) | 2 (2)
High alkaline phosphatase (Investigations) | 2 (7)
High ALT (Investigations) | 3 (9)
High AST (Investigations) | 5 (14)
Hyperbilirubinemia (Investigations) | 5 (14)
Hyperglycemia (Investigations) | 3 (11)
Hypertension (Cardiac disorders) | 2 (2)
Hypoalbuminemia (Investigations) | 2 (5)
Hypocalcemia (Investigations) | 3 (7)
Hypokalemia (Investigations) | 3 (7)
Hypophosphatemia (Investigations) | 2 (3)
Hypotension (Cardiac disorders) | 7 (23)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Incontinence (Musculoskeletal and connective tissue disorders) | 3 (7)
Infection (Infections and infestations) | 5 (8)
Insomnia (Nervous system disorders) | 2 (2)
Leukopenia (Investigations) | 8 (42)
Lightheadedness (Cardiac disorders) | 4 (5)
Lymphopenia (Investigations) | 4 (26)
Mucositis (Gastrointestinal disorders) | 2 (7)
Nausea (Gastrointestinal disorders) | 6 (18)
Neuropathy (Nervous system disorders) | 9 (19)
Neutropenia (Investigations) | 5 (17)
Pain - general (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain - abdomen (Musculoskeletal and connective tissue disorders) | 7 (12)
Pain - back (Musculoskeletal and connective tissue disorders) | 9 (15)
Pain - chest (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain - foot (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - hip (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - leg (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain - neck (Musculoskeletal and connective tissue disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Renal failure (Renal and urinary disorders) | 2 (2)
Somnolence (Nervous system disorders) | 2 (3)
Sweating (Skin and subcutaneous tissue disorders) | 4 (4)
Tachycardia (Cardiac disorders) | 2 (3)
Thrombocytopenia (Investigations) | 6 (36)
Thrush (Infections and infestations) | 4 (5)
Transfusion reaction (Immune system disorders) | 3 (4)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2)
Vaginal bleeding (Reproductive system and breast disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (20)
Weakness (Nervous system disorders) | 3 (11)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Xerostomia (Gastrointestinal disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes